CLINICAL TRIAL: NCT02369783
Title: Screening for Social Weaknesses and Coordination Course of Cancer Patients: A New Approach by an Expert System IT
Brief Title: Screening for Social Weaknesses and Coordination Course of Cancer Patients
Acronym: DEFCOCANCERO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2014-05
Record Dates: First submitted 2015-02-06; First posted 2015-02-24 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Questionnaire and interview (Experimental): The patient complete the questionnaire on the tablet to better know their social situation and any difficulties. Then, he will be interview during thirty minutes with a social worker and a nurse navigator. At the end of this intervention we will be offered to the patient monitoring and appropriate resources to its situation.
  Interventions: Other: Questionnaire and interview

INTERVENTIONS:
Other: Questionnaire and interview — The aim is to detect social fragility.

SUMMARY:
The main objective of the study is to validate a methodology with Psychometric tool to measure levels of patients social fragility.

This tool will be dematerialized on a tablet. The answers will be then processed by a decision support algorithm, which automatically send an alert to detection of social fragility of the patient to the nurse navigators.

ELIGIBILITY:
Inclusion Criteria:

* All new patients enter ICLN for a diagnosis of cancer
* Patients who can read French or patients who can not read French, but accepting the translation by a close friend or family
* Patient having signed a free and informed consent

Exclusion Criteria:

* Refusal of participation, major patients protected under guardianship.
* Patient can not read French without possibility of translation by a close friend or family

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Questionnaire validity | 1 hour
  Outcomes are content validity by expert judges method, appearance validity through a consensus, construct validity through exploratory factor analysis, discriminant validity in relation to the social fragility through univariate analysis, internal validity through factor analysis

CONTACTS AND LOCATIONS:
Overall Officials: Franck Chauvin, PhD-MD, Study Director — INSTITUT DE CANCEROLOGIE DE LA LOIRE
Locations (1):
- Institut de Cancerologie de la Loire, Saint-Priest-en-Jarez, France